CLINICAL TRIAL: NCT04899011
Title: Taste Disturbance After Middle Ear Surgery: Frequency, Duration, Influence of Chorda Tympani Injury and Quality of Life
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21IUFC01
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Ear Middle Problems
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Middle ear surgery
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire about taste and salivary disturbance before surgery, 10 days, 4 months and 1 year after surgery.
  Questionnaires include characteristics of taste disturbance, and specific impact on quality of life.

SUMMARY:
Chorda tympani nerve (CTN), is a branch of nerve VII, and has two componants: taste sensation from the anterior two thirds of the tongue and salivary secretion from submandibular and sublingual salivary glands.

CTN go throw middle ear between malleus and incus. Due to it anatomic localization, CTN is frequently damage during otologic surgery.

Taste disturbance after middle ear surgery has been describe in literature but results of the various studies are very heterogenous. Moreover, there is no consensus to preserved or sacrificed a traumatize CTN.

We will use questionnaire to evaluate frequency, duration and characteristics of taste disturbance after ear surgery and the impact on the quality of life for those with symptoms.

We will evaluate the Influence of type of CTN injury on taste disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing middle ear surgery
* Acceptation to participate
* under 18 years old, parental authorization.

Exclusion Criteria:

* Taste disturbance before surgery
* Patients with guardianship or tutelage measure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with middle ear surgery
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Frequency, duration and characteristics of taste and salivary disturbance after middle ear surgery and impact on quality of life. | 1 year
  Taste and salivary disturbance will be measure with questionnaire before and during 1 year after middle ear surgery

SECONDARY OUTCOMES:
Influence of CTN injury type: stretch versus sectionned, influence of otologic desease | 1 day
  Measure with surgeon questionnaire
Influence of use between endoscope or microscope surgery | 1 day
  Measure with surgeon questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GUEVARA, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No